CLINICAL TRIAL: NCT00656565
Title: Inspiratory Flow Rates and Volumes in Subjects With Bronchiectasis Using Low and High Resistance Dry Powder Inhaler Devices
Brief Title: Inspiratory Flow and Volumes in Bronchiectatics
Status: Completed | Type: Observational
Sponsor: Syntara (Industry)
Responsible Party: Dr Sandra Anderson, Royal Prince Alfred Hospital
Other Study IDs: DPM-OSM-402
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Bronchiectasis
Keywords: measure inspiratory spirometry with dry powder inhaler device in series with the spirometer
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: subjects with bronchiectasis

SUMMARY:
Adequate administration of drugs via dry powder inhalers is dependent on adequate inspiratory flow rates and volumes. These vary according to the device being used and its resistance. The dry powder inhaler device under investigation is a device approved by the Therapeutic Goods Administration (ARTG no. 196255) for use with dry powder mannitol. Dry powder mannitol is currently being investigated as a treatment for bronchiectasis. We wish to measure the inspiratory flow characteristics of both the low and high resistance devices amongst a group of subjects with bronchiectasis.

We propose that the majority of subjects investigated with varying lung function will achieve adequate flow during a controlled inspiration.

ELIGIBILITY:
Inclusion Criteria:

* non-cf bronchiectasis
* aged 18-80 inclusive
* FEV1 greater or equal to 50% predicted and greater or equal to 1L

Exclusion Criteria:

* uncontrolled asthma
* CF bronchiectasis
* have any condition for which spirometry measurement would be contraindicated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects aged 18-80 years, with bronchiectasis and FEV1 greater or equal to 50% predicted and greater or equal to 1L
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
inspiratory flow | single visit

SECONDARY OUTCOMES:
inspiratory volume | single visit

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia